CLINICAL TRIAL: NCT05680207
Title: The Effect of Empowerment Training on Type 2 Diabetes Patients on Empowerment Levels and Clinical Findings: A Randomized Controlled Trial
Brief Title: Empowerment Training on Type 2 Diabetes Patients on Empowerment Levels and Clinical Findings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Muzelfe BIYIK, Master of Science, Kutahya Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DM Training
Record Dates: First submitted 2022-12-20; First posted 2023-01-11 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Diabetes Mellitus, Type 2; Empowerment; Patient Empowerment
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Empowerment; Patient Participation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): Type 2 Diabetes Mellitus patients who received a empowerment training program for 6 weeks, 2 hours a week
  Interventions: Behavioral: Diabetes self- management education (DSME) program
- Control group (No Intervention): Type 2 Diabetes Mellitus patients who did not receive a empowerment training program

INTERVENTIONS:
Behavioral: Diabetes self- management education (DSME) program — We offered a two-hour course each week, comprising of two sessions of lectures (40 minutes each), two breaks (10 min each) and interactive session (20 min). In the interactive session, patients could communicate with each other in groups or raise any questions to the investigators.
  Arms: Intervention group

SUMMARY:
In this study, the effect of nurse-led empowerment training given to patients with Type 2 Diabetes on clinical findings and empowerment behaviors will be investigated.

DETAILED DESCRIPTION:
The research is a randomized controlled design research that includes a pre-test/post-test design. The primary outcome expected in the research; change in empowerment behaviors as a result of the training given; secondary outcomes are changes in clinical findings.

The research universe; All Type 2 diabetes patients who applied to the endocrinology polyclinic of a private hospital in Eskisehir city center between March-July 2019 consisted of. In the study, the sample was randomly selected, and it was aimed to reach all patients with Type 2 diabetes who were 18 years of age and older, with a diagnosis period of one year or more.

In the study, patients were randomly assigned to the intervention group, which included 6 weeks of training, or to the control group, which was on a 6-week waiting list. It used a question-based format to address the educational, behavioral, and psychosocial needs of patients within the scope of a 12-hour empowerment program that lasted for 6 weeks, 2 hours a week.

Education (DSMS (Developing Empowerment-Based Diabetes Self-Management Support)) is planned as stated literature.

Purpose of education: Empowerment as a philosophy of care emphasizes a collaborative approach to facilitating behavior change for patients themselves. Empowerment approach; Goal setting is a five-step process that provides patients with the knowledge and clarity they need to develop and achieve their diabetes and lifestyle goals. The first two steps are to identify the problem and identify patients' beliefs, thoughts, and feelings that may support or hinder their efforts. The third step is to determine the long-term goals expected from patients. In this step, patients are then expected to make a behavioral change that will help them achieve their long-term goals. The last step is for patients to evaluate their efforts and determine what they have learned in the process. Empowerment training was determined within the framework of this process.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Type 2 Diabetes Mellitus diagnosed more than 1 year ago

Exclusion Criteria:

* Mental retardation
* Dementia
* Deafness
* Blindness
* Psychiatric illness
* Steroid use

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
improvement in The Diabetes Empowerment Scale scores | 3 months
  The Diabetes Empowerment Scale (DES-28) questionnaires consist of 28 items with 3 subscales, with each item rated along a 5-point Likert scale (1 = strongly disagree, 2 = disagree, 3 = neutral, 4 = agree, 5 = strongly agree). The range of score was divided in three subgroups as low (28-65 scores), middle (66-103) and high (104-140).
  All items have been scored so that a higher value indicates stronger empowerment.

SECONDARY OUTCOMES:
improvement in HbA1c levels | 6 months
  decrease in HbA1c (mmol/mol)
improvement in fasting glucose | 6 months
  decrease in fasting glucose (mmol/L)
improvement in low density lipoprotein | 6 months
  decrease in low density lipoprotein (mmol/L)
improvement in triglyceride | 6 months
  decrease in triglyceride (mmol/L)

CONTACTS AND LOCATIONS:
Overall Officials: müzelfe bıyık, Ms, Study Chair — Eskişehir Osmangazi University
Locations (1):
- Acıbadem Hospital, Eskişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Messina R, Rucci P, Sturt J, Mancini T, Fantini MP. Assessing self-efficacy in type 2 diabetes management: validation of the Italian version of the Diabetes Management Self-Efficacy Scale (IT-DMSES). Health Qual Life Outcomes. 2018 Apr 23;16(1):71. doi: 10.1186/s12955-018-0901-3. PMID 29685153